CLINICAL TRIAL: NCT05758753
Title: The Efficacy of Quantitative Sensory Test (QST) in Assessing Corneal Nerve Functions in Patients With Ocular Surface Diseases
Brief Title: QST for Corneal Nerve Function
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving institution. USF will likely resume study activity but TMC is no longer conitinuing study activity.
Sponsor: Tufts Medical Center (Other)
Collaborators: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002510
Record Dates: First submitted 2022-09-06; First posted 2023-03-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Corneal Disease; Neuropathy; Dry Eye Disease; Neurotrophic Keratitis
Keywords: Quantitative Sensory Test
MeSH Terms: conditions — Corneal Diseases; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage I Neurotrophic Keratopathy (Experimental): Clinical findings of corneal hyperplasia and irregularity, scattered small facets of dried epithelium, decreased nerve density as assessed by in vivo confocal microscopy (IVCM), and decreased corneal sensation.
  Interventions: Device: Quantitative Sensory Test
- Stage II Neurotrophic Keratopathy (Experimental): Clinical findings of corneal epithelial defect with smooth and rolled edges, decreased nerve density as assessed by in vivo confocal microscopy (IVCM), and decreased corneal sensation.
  Interventions: Device: Quantitative Sensory Test
- Dry Eye Disease (Experimental): Symptoms of dry eye disease for at least 3 months, supported by clinical finding of decreased tear film break-up time or ocular surface staining. Normal corneal sensation.
  Interventions: Device: Quantitative Sensory Test
- Healthy Individuals (Experimental): Absence of any ocular symptoms, absence of surface findings (including corneal or conjunctival staining, corneal scar or surgical wound), and normal corneal sensation.
  Interventions: Device: Quantitative Sensory Test

INTERVENTIONS:
Device: Quantitative Sensory Test — Quantitative Sensory Test (Medoc Ltd, Israel), QST is a non-invasive neurophysiological method that refers to a group of procedures that assess the perceptual responses to systematically applied and quantifiable sensory stimuli (modalities including heat, cold and vibration) for the purpose of characterizing somatosensory function or dysfunction. For this test, subjects will be seated comfortably on a chair in a quiet room, or laying supine in a horizontal examination chair, with ambient temperature of 24-25◦ C. Medial upper eyelid; just below the supraorbital notch, nasolacrimal sac area; 4-5 mm medial to nasal cantus, and non-dominant forearm will be used as test sites. Patients will be instructed in detail of the nature of the test and the need to react attentively and promptly to change in temperatures.

SUMMARY:
This study is designed to learn more about the impact different types of stimuli, such as heat, cold and vibration, can have on ocular pain response. This is called quantitative sensory testing (QST). Most procedures being performed in this study, except the QST, are standard of care which means they are performed during the participant's routine eye examination.

DETAILED DESCRIPTION:
Quantitative Sensory Test (QST) is a non-invasive neurophysiological method that refers to a group of procedures that assess the perceptual responses to systematically applied and quantifiable sensory stimuli for the purpose of characterizing somatosensory function or dysfunction.

In this study, we propose to evaluate corneal nerve functions in patients with corneal nerve abnormalities by QST and correlate the nerve functions with symptoms, clinical signs and nerve morphology detected by In-Vivo Confocal Microscopy (IVCM). Identification of corneal nerve functions and correlations with other findings may help us to understand underlying pathological mechanisms of the disease and may guide us toward new treatment targets.

We hypothesize that, QST may provide us detailed information about corneal nerve function alterations and may correlate with morphological nerve changes detected by IVCM.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Stage I Neurotrophic Keratopathy (NK)

1. Clinical findings of Stage I NK
2. Decreased nerve density by IVCM
3. Decreased corneal sensation

Group 2: Stage II NK

1. Clinical findings of Stage II NK
2. Decreased nerve density by IVCM
3. Decreased corneal sensation

Group 3: Dry Eye Disease (DED)

1. Symptoms of DED at least 3 months
2. Presence of at least one of the following DED signs; tear film break-up time lower than 7, ocular surface staining more than +1 based on NIH scale
3. Normal or mildly effected corneal sensation

Group 4: Healthy Individuals

1. Absence of any ocular surface symptoms
2. Absence of ocular surface findings
3. Transparent and clear cornea
4. Normal corneal sensation

Group 5: NCP

1. Presence of neuropathic symptoms AND
2. Symptoms out of proportion to clinical findings AND
3. Nerve abnormalities detected by in vivo confocal microscopy

Exclusion Criteria:

1. History of diabetes
2. History of ocular surgery, corneal infection, or corneal injury within the last 3 months
3. Systemic regular anti-inflammatory and/or steroid and/or immune-modulatory therapy in the last 3 months
4. Active ocular allergies
5. Any major psychiatric illness including bipolar, psychosis, obsessive-compulsive disorder and major depression
6. Pregnancy
7. History of surgery within the last 3 months
8. History of , sarcoidosis, GVHD or collagen vascular disease
9. Allergic to benzalkonium chloride "BAK" (an eye-drop preservative)
10. Concurrent enrollment in other studies that in the opinion of the investigator will interfere with the results of this study
11. Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Thermal stimulus response to QST on site of trigeminal nerve first branch, as assessed by cold detection threshold (CDT) and hot detection threshold (HDT) | From visit 1 up to 4 weeks
  Cold and heat sensation thresholds will be evaluated by placing a 16 mm x 16 mm probe over the skin on the site to be tested, and an average of 3 reading while be taken for each stimuli. Participants will receive successive ramps of gradually decreasing or increasing temperature, starting from a resting neutral temperature of 32°C. Participants will be instructed to press a response button when a thermal sensation (either cold or warm) is perceived.
Mechanical stimulus response to QST on site of trigeminal nerve first branch, as assessed by vibration detection threshold (VDT) | From visit 1 up to 4 weeks
  Vibration sensation threshold will be evaluated by placing a 16 mm x 16 mm probe over the skin on the site to be tested, and an average of 3 reading while be taken. Participants will receive successive ramps of gradually decreasing or increasing vibration, starting from. Participants will be instructed to press a response button when a mechanical sensation is perceived.
Differences in thermal stimulus pain threshold across the 4 study arms | From visit 1 up to 4 weeks
  Cold pain threshold (CPT) and heat pain threshold (HPT) will be measured by asking participants to press a response button when they first feel a pain or discomfort from probe on QST testing
Differences in mechanical stimulus pain threshold across the 4 study arms | From visit 1 up to 4 weeks
  Vibration pain threshold (VPT) will be measured by asking participants to press a response button when they first feel a pain or discomfort from vibration probe on QST testing

SECONDARY OUTCOMES:
To correlate the QST responses with morphological changes of corneal nerves detected by IVCM | From visit 1 up to 4 weeks
  In vivo confocal microscopy (IVCM) imaging will be performed to observe for any morphological nerve changes; such as decreased nerve density, nerve tortuosity presence of microneuromas.
To correlate symptom severity as assessed by the Ocular Surface Disease Index (OSDI), to stimulus response across the 4 interventional arms. | From visit 1 up to 4 weeks
  Ocular Surface Disease Index (OSDI) questionnaire A 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning. The 12 items of the OSDI questionnaire are graded on a scale of 0 to 4, where 0 indicates none of the time; 1, some of the time; 2, half of the time; 3, most of the time; and 4, all of the time. The total OSDI score is then calculated on the basis of the following formula: OSDI= [(sum of scores for all questions answered) x 100]/[(total number of questions answered) x 4]. Higher OSDI scores represent greater severity of symptoms.
To compare QST response differences between trigeminal nerve first branch and forearm in patients. | From visit 1 up to 4 weeks
  Measurement of stimuli detection thresholds, pain thresholds and pain ranges for different stimuli (cold, heat and vibration) type in study groups at 3 different periocular sites (just below supraorbital notch, lateral canthus, inferior orbital bone; 1 cm lateral of medial canthus) and non-dominant hand hypothenar eminence (as a reference site)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No